CLINICAL TRIAL: NCT03136822
Title: Clinical Evaluation of the Wound Dressing Impregnated With Microparticules (DERMALIX) on Diabetic Foot Ulcers
Brief Title: DERMALIX Efficacy on Diabetic Foot Ulcers
Acronym: DERMAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dermis Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DERMAN
Record Dates: First submitted 2017-04-28; First posted 2017-05-02 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Diabetic Foot; Diabetic Foot Ulcer
Keywords: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Open label, controlled, randomised, parallel arm study
Who Masked: Outcomes Assessor
Masking Description: The wound will be assessed by Pathologists who are masked for treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Standard dressing
  Interventions: Other: Standard Dressing
- Treatment (Experimental): Standard dressing + Wound dressing (DERMALIX)
  Interventions: Other: Standard Dressing; Device: DERMALIX

INTERVENTIONS:
Other: Standard Dressing — Standard dressing is applied for treatment of diabetic foot ulcers
Device: DERMALIX — DERMALIX, a class III Medical Device will be applied in addition to standard dressing
  Arms: Treatment

SUMMARY:
(DERMALIX) (Patent number: PCT/TR2014/000251) is a bioactive wound dressing that was developed by Ege University School of Pharmacy Department of Pharmaceutical Technology. This dressing has been categorised as Class III medical device. This clinical study will be conducted in patients with diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 Patients diagnosed with diabetic foot ulcers
* Class I and II according to Wagner classification
* No infections confirmed with culture test
* No osteomyelitis and gangrene in the foot
* HbA1c values ≤ % 7.5
* Not active smoker
* No planned treatment of hyperbaric oxygen
* Patients who give consent for the study

Exclusion Criteria:

* Patients with diabetic foot ulcer of class 3,4 and 5 according to Wagner classification
* Patients who are pregnant or breast-feeding or female who are in reproductive age applying no preservative method
* Patients who have mental conditions that lead to difficulties in comprehension
* Patients who may have compliance issues
* Patients who have been included to another interventional study with drug or medical device

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Recovery of the wound 100% | 1 month
  The wound will be completely recovered

SECONDARY OUTCOMES:
Recovery of the wound 80% | 1 month
  The wound will be recovered by 80%

CONTACTS AND LOCATIONS:
Overall Officials: Sevki Cetinkalp, Prof, Principal Investigator — Ege University School of Medicine
Locations (1):
- Ege University School of Medicine, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No